CLINICAL TRIAL: NCT00532753
Title: Evaluating the Hunger Project's Scaling-up of Epicenter Strategy in Ghana
Brief Title: Evaluating the Hunger Project in Ghana
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of California, Berkeley (Other)
Collaborators: The Robertson Foundation (Other)
Responsible Party: Dr. David I. Levine, UC Berkeley
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CPHS Protocol #2007-4-42
Record Dates: First submitted 2007-09-18; First posted 2007-09-20 (Estimated); Last update posted 2008-08-04 (Estimated); Status verified 2008-07

CONDITIONS: To Better Understand How Epicenter's (Which House Education, Health and Finance Centers in Ghana) Increase Individual's Sense of Empowerment.
Keywords: empowerment; health; education
MeSH Terms: conditions — Empowerment

INTERVENTIONS:
Behavioral: Community Empowerment

SUMMARY:
The Hunger Project/Epicenter strategy is a community based development strategy that will positively affect health, education, empowerment, and consumption.

DETAILED DESCRIPTION:
The investigators propose a randomized controlled design that will measure how The Hunger Projects' intervention affects the lives of Ghanaians. A pre-intervention baseline survey of approximately 4,000 households with over 20,000 individuals and two follow-up surveys of the same households will be conducted over the ten year experimental period.

ELIGIBILITY:
Inclusion Criteria:

* The subject population will be individuals and households from communities in the Eastern Region of Ghana.

Exclusion Criteria:

* Only exclusion criteria is that households outside of the Eastern region of Ghana will not be surveyed

Sex: All
Age Groups: Child, Adult, Older Adult
Enrollment: 20000 (Estimated)
Dates: Start 2007-08; Primary Completion 2010-08; Study Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
Increased sense of empowerment

SECONDARY OUTCOMES:
Increased health, education, and consumption outcomes and increase in the number of public goods

CONTACTS AND LOCATIONS:
Overall Officials: David Levine, PhD Econ, Principal Investigator — University of California at Berkeley
Locations (1):
- Ghana Hunger Project, Several, Eastern Region, Ghana